CLINICAL TRIAL: NCT05307211
Title: Evaluation of the Effect of Stabilization Exercises on Interlaminar Epidural Steroid Injection Treatment Results in Cervical Radiculopathy
Brief Title: Are Stabilization Exercises Effective After Epidural Steroid Injection in Patients With Cervical Radiculopathy?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 04.03.2022.357
Record Dates: First submitted 2022-03-22; First posted 2022-04-01 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Pain, Neck; Cervical Radiculopathy; Pain, Radiating
Keywords: Pain; cervical radiculopathy; cervical interlaminar epidural steroid injection; stabilization exercises
MeSH Terms: conditions — Neck Pain; Radiculopathy; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GROUP 1 (CIESI Only) (Active Comparator): Only interlaminar epidural steroid injection will be administered to patients in this arm with the same method as in the other arms (one session, week 0). Staying active will be the only recommendation, and no exercise prescription will be provided.
  Interventions: Procedure: Cervical Interlaminar Epidural Steroid Injection
- GROUP 2 (CIESI plus NECK STABILIZATION EXERCISES) (Experimental): After the interlaminar epidural steroid injection, the patients will be taken to an exercise program in the physical therapy unit, in the company of a physiotherapist, within 24 hours, within 72 hours at the latest.
  Interventions: Procedure: Cervical Interlaminar Epidural Steroid Injection; Other: Neck Stabilization Exercises
- GROUP 3 ( CIESI plus NECK and SCAPULAR STABILIZATION EXERCISES) (Experimental): After the interlaminar epidural steroid injection, the patients will be taken to an exercise program in the physical therapy unit, in the company of a physiotherapist, within 24 hours, within 72 hours at the latest.
  Interventions: Procedure: Cervical Interlaminar Epidural Steroid Injection; Other: Neck and Scapular Stabilization Exercises

INTERVENTIONS:
Procedure: Cervical Interlaminar Epidural Steroid Injection — Fluoroscopy-guided cervical interlaminar epidural steroid injection will be administered to patients with chronic neck pain due to cervical disc herniation. The injection area is cleaned 3 times with an antiseptic solution and covered with a sterile cloth. Local anesthesia with 2 ccs 3% prilocaine will be applied to the skin and subcutaneous tissues in the area of interest. Under fluoroscopy guidance, the needle is advanced into the C7-T1 intervertebral disc level. With the help of the loss of resistance technique, it is understood that the needle is in the epidural space, and second control is provided by administering contrast material. After the confirmation of needle place is done, a mixture of 12 mg dexamethasone, 1 cc 2% lidocaine, 1 cc saline is injected. The patient is taken to the restroom after the procedure and followed up for any complications.
Other: Neck Stabilization Exercises — The physiotherapist will design an exercise protocol for neck stabilization. Each exercise will be applied three days a week throughout a 4-week program, accompanied by a physiotherapist, and will begin with 7 to 10 repetitions at first, increasing to 10 to 15 repetitions in the following weeks, taking into account the patient's condition. After the physiotherapist-assisted exercises are completed, the protocol will continue as home-based exercises until the assessments are completed.
  Arms: GROUP 2 (CIESI plus NECK STABILIZATION EXERCISES)
Other: Neck and Scapular Stabilization Exercises — The physiotherapist will design an exercise protocol for neck and scapular stabilization. Each exercise will be applied three days a week throughout a 4-week program, accompanied by a physiotherapist, and will begin with 7 to 10 repetitions at first, increasing to 10 to 15 repetitions in the following weeks, taking into account the patient's condition. After the physiotherapist-assisted exercises are completed, the protocol will continue as home-based exercises until the assessments are completed.
  Arms: GROUP 3 ( CIESI plus NECK and SCAPULAR STABILIZATION EXERCISES)

SUMMARY:
Cervical radiculopathy was first described in 1943 by researchers named Semmes and Murphy, years later than lumbosacral radiculopathy. It is a neurological condition caused by dysfunction in the cervical spinal nerves, nerve roots, or both. This compression occurs as a result of disc herniation, spondylosis, trauma, spinal tumors, etc. As the first symptom, it manifests as pain. When pain radiates from the neck to the shoulder and arm and is accompanied by sensory complaints and motor weakness, cervical radiculopathy should be suspected. It is a significant cause of morbidity and disability in both men and women, and it occurs in middle age. As a result, clinicians must quickly diagnose and determine the best treatment method. The majority of the information in the literature on the incidence of cervical radiculopathy is based on the findings of a large population-based study conducted between 1976 and 1990 by the Mayo Clinic in Rochester, Minnesota. The incidence rate of cervical radiculopathy was reported to be 83.2 per 100,000 per year in this study, which included 561 cases. The primary goals of treatment are to alleviate pain, restore neurological function, and prevent a recurrence. According to the literature, cervical radiculopathy recurs at a rate of 31.7%, and 26% of them go to surgery. Treatment options vary depending on whether the symptoms are acute or chronic and their severity. In the treatment of cervical radiculopathy, either conservative (non-operative) or surgical treatments are used. In patients with chronic neck pain with or without radiculopathy, a cervical epidural steroid injection is one of the most frequently used interventional therapeutic options. Chronic neck pain or radicular pain caused by disc herniation, spinal stenosis, or discogenic pain can also be treated with cervical epidural injections. Cervical stability training is an exercise program that is used to strengthen the cervical spine, relieve pain, and improve functionality. Changes in dynamic scapula stabilization are observed in patients with chronic neck pain. The scapula connects the neck and shoulder, so it plays an important role in stabilizing the neck and shoulder complex. Because of the interaction between the neck and the scapula, scapular stability becomes more important in these patients.

DETAILED DESCRIPTION:
Many studies in the literature separately investigate the effectiveness of Cervical Interlaminar Epidural Steroid Injection (CIESI) in radiculopathy due to cervical disc herniation or the effectiveness of stabilization exercises and physical therapy modalities in these patients. However, there have been no studies on the effectiveness of post-injection exercise training as far as we are aware. Our study aims to investigate the benefit of stabilization exercises after interlaminar epidural steroid injection in patients with radiculopathy caused by cervical disc herniation, add a new study to the literature, and guide future research.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65
* Cervical radiculopathy has caused neck and arm pain for at least three months.
* Sign a consent form and volunteer to take part in the study.

Exclusion Criteria:

* Previous surgical/interventional procedure for the cervical region
* Presence of other musculoskeletal disorders (such as lateral epicondylitis, tendinitis, entrapment neuropathy) that may cause diagnostic confusion in terms of pain pattern and localization
* Signs of trauma, fracture, malignancy, or active infection
* Rheumatological (RA, AS, etc.), endocrinological (such as osteoporosis, Paget's disease), or another systemic disease that may change the anatomical or physiological structure of the relevant regions Presence of coagulopathy
* History of whiplash injury, cervical spinal stenosis, cervical spondylosis
* Being pregnant and breastfeeding
* Presence of mental deterioration or psychiatric/neurological disease that can affect the flow of the study.
* Having a history of allergic reactions to the injectables that will be used.
* Presence of cardiopulmonary disease that may lead to exercise intolerance (heart failure, chronic obstructive pulmonary disease, etc.)
* Failure to implement the exercise program regularly.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-04-29 (Actual)

PRIMARY OUTCOMES:
Change of pain severity from baseline to each checkpoints | from pre-interventional time to post-interventional 1st hour, 1st month, 3rd month
  The numerical rating scale (NRS) is widely used in research and clinical settings to represent pain intensity. NRS is defined as 0 for the absence of pain and 10 as the worst possible pain. The NRS is moderately reliable and has a clinically important difference (CID) value of 1.0.

SECONDARY OUTCOMES:
Change of functionality from baseline to each checkpoints | from pre-interventional time to post-interventional 1st month, 3rd month
  The Neck Disability Index (NDI) is a validated 10-item questionnaire that measures a patient's self-reported disability due to neck pain. The score ranges from 0 (no disability) to 100 (completely disabled). The minimum detectable change (MDC) for patients with cervical radiculopathy is 10 points, and the clinically important difference (CID) is 14 points.
Change of life quality from baseline to each checkpoints | from pre-interventional time to post-interventional 1st month, 3rd month
  Short Form-12 (SF-12) is a scale that was developed in 1994 to evaluate the quality of life for the last four weeks without focusing on a specific age and disease group. It consists of 12 questions, all selected from the SF-36 Health Questionnaire. SF-12 consists of physical functionality, physical role, pain, general health, emotional role, mental health, social functionality, and vitality sub-components.

CONTACTS AND LOCATIONS:
Overall Officials: Savaş Şencan, MD, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Faculty of Medicine, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tayboga UI, Olgun Y, Gunduz OH, Sencan S. Are Stabilisation Exercises Effective After Epidural Steroid Injection in Patients With Cervical Radiculopathy? A Prospective Randomised Controlled Trial. Eur J Pain. 2025 Feb;29(2):e4777. doi: 10.1002/ejp.4777. PMID 39779455